CLINICAL TRIAL: NCT05014750
Title: Zhongshan Hospital, Fudan University
Brief Title: Frailty of Elderly With Valvular Heart Disease and the Short Term Adverse Events
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Frailty Study 01
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-08

CONDITIONS: Frailty; Elderly; Valvular Heart Disease
MeSH Terms: conditions — Frailty; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None intervention — There is no intervention included in this study.

SUMMARY:
Despite the rapid development of medical and nursing technology, the prognosis of valvular heart disease has been greatly improved. However, compared with young patients, the mortality and adverse event rate of elderly patients with valvular heart disease are still high, surgical complications are more frequent and hospitalization time is longer. The complexity of valvular heart disease and the poor prognosis in the elderly forces us to continue to look for other potential prognostic factors. In addition to the adverse outcomes caused by disease factors, elderly patients with valvular heart disease also have the gradual decline of physiological and psychological reserve function caused by age factors. These adverse outcomes include osteopenia, disability, prolonged hospitalization and even death are all closely related to frailty. Frailty is 'a biologic syndrome of decreased reserve and resistance to stressors, resulting from cumulative declines across multiple physiologic systems, and causing vulnerability to adverse outcomes. The essence of frailty is the decline of individual resistance, which eventually leads to the increase of individual brittleness and susceptibility to adverse health outcomes. At present, the research in the field of elderly vulnerable groups of cardiovascular disease in China started late, mostly focusing on the study of pathological mechanism, the introduction of evaluation tools, conceptual analysis and so on. Almost all of the existing studies are about the debilitation status of elderly patients with heart valve disease, and most of them mainly try to find the influencing factors of debilitation from the aspects of patients' physical diseases, ignoring the impact of factors such as the mental health status of the elderly on debilitation, there are few reports of short-term adverse events in elderly patients with valvular heart disease. This study will analyze the influencing factors of the weakness of elderly patients with valvular diseases from the multi-dimensional aspects of demographic data, physical diseases, psychology and society, and track the short-term prognosis of patients with death, fall and unconventional rehospitalization, so as to provide a research basis for relevant research in the future.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years;
* Willing to continue to participate in this study;
* Diagnosed as valvular heart disease

Exclusion Criteria:

* suffering from other irreversible serious diseases;
* with severe mental disorders;
* cannot accept frailty assessment due to treatment needs and other factors.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients with valvular heart disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Death | One year after discharge
  All-cause death
Falls | One year after discharge
  Falls
Rehospitalization | One year after discharge
  Unplanned rehospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No